CLINICAL TRIAL: NCT07247474
Title: Characterizing the Evolution of Neonatal Lung Disease Throughout Infancy and Childhood Using Electrical Impedance Tomography: A Pilot Study
Brief Title: Triple EIT (Electrical Impedance Tomography)
Status: Recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: Colorado State University (Other)
Responsible Party: Sponsor
Other Study IDs: 25-1298
Record Dates: First submitted 2025-11-11; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Neonates and Preterm Infants; Cardiopulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Cardiopulmonary disease: Have evidence of cardiopulmonary disease including, but not limited to:
  * Post-prematurity respiratory disease
  * Congenital diaphragmatic hernia
  * Pulmonary hypertension
  * Congenital heart disease
  * Respiratory failure
  * Neuromuscular disease
  * Developmental or congenital lung disease
  May be imaged with two machines
  Interventions: Device: Electrical impedance tomography (EIT)
- Control: matched healthy controls with no cardiopulmonary disease
  Interventions: Device: Electrical impedance tomography (EIT)

INTERVENTIONS:
Device: Electrical impedance tomography (EIT) — Electrical impedance tomography (EIT) is a noninvasive and non-ionizing imaging technique that describes lung ventilation and perfusion

SUMMARY:
This study plans to learn more about ways to look at participant's lungs using new machines called Electrical Impedance Tomography (EIT). The EIT does not use harmful radiation like CT or x-ray. It is read through electrodes like using EKG reading heartbeats.

The investigators want to compare the results of patients who have chronic respiratory disease to patients without chronic respiratory disease to learn more about lung structure and composition.

ELIGIBILITY:
Inclusion Criteria:

* 2 weeks to 25 years of age
* evidence of cardiopulmonary disease including, but not limited to:

  1. Post-prematurity respiratory disease
  2. Congenital diaphragmatic hernia
  3. Pulmonary Hypertension
  4. Congenital heart disease
  5. Respiratory failure
  6. Neuromuscular Disease
  7. Developmental or congenital lung disease

OR matched healthy controls (born at term gestation (>36 weeks gestational age) with no cardiopulmonary disease)

Exclusion Criteria:

* <2 weeks of age
* Anything that interferes with lead placement on the chest wall (such as, dermatologic conditions, multiple chest tubes, anatomic abnormality, or large dressings that cannot be moved)
* No informed consent
* Pregnant or lactating
* Pacemaker or other metal intrathoracic surgical implant (causes noise in the data)

Ages: 2 Weeks to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children's Hospital Colorado
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2028-11 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
EIT Imaging Maps that provide information about regional ventilation and perfusion of the lung | 4 hours
  These images will be analyzed both visually for qualitative abnormalities and through quantitative pixel analysis that can provide information regarding lung volume, blood volume, and changes in either based on respiratory cycle, cardiac cycle, or intervention. Areas of low ventilation (atelectasis and consolidation) will be identified.

SECONDARY OUTCOMES:
Regional Conductivity Due to Ventilation | 4 hours
  This is a qualitative aim and will summarize EIT images pictorially. Pixel densities will be evaluated for normality and summarized as mean (SD) or median (interquartile range). EIT images will be qualitatively compared between cases and controls. Outcome metrics may be generated to measure things such as ventilation heterogeneity
Regional Conductivity Due to Perfusion | 4 hours
  This is a qualitative and quantitative aim that will only be performed using the ACT5 EIT system. Results will qualitatively compare EIT images with CXR and CT scan images when available. Images will be displayed side by side and interpreted by both the clinician and the EIT study staff. Various summary measures of EIT outcomes will be calculated including pixel heterogeneity, summary changes over tidal breath and variation between tidal peaks. Pearson and Spearman correlation will be calculated between summary EIT outcomes and continuous primary clinical values. Linear and logistic regression will be used to estimate associations (with 95% CI) between EIT measures and clinical outcomes. Summary data will be presented in tables and figures using basic descriptive statistics stratified by study group.
Comparison of Ventilation and Perfusion Ratio | 4 hours
  In participants with both ventilation and perfusion metrics from the ACT5 EIT system, a regional comparison of ventilation and perfusion will be generated. These values will indicate whether a segment of the lung has relatively more or less ventilation or perfusion.

CONTACTS AND LOCATIONS:
Overall Officials: Katelyn Enzer, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No